CLINICAL TRIAL: NCT04517188
Title: A Phase 4 Study to Evaluate Nasopharyngeal SARS-CoV-2 Viral Shedding After Halodine Nasal Antiseptic in Patients With COVID-19
Brief Title: Halodine Nasal Antiseptic in Patients With COVID-19
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Halodine LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HDN-N02-COV24A
Record Dates: First submitted 2020-08-15; First posted 2020-08-18 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: SARS-CoV-2 Infection
Keywords: Nasopharyngeal SARS-CoV-2 Viral Load
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Halodine Nasal Antiseptic (Experimental): Povidone-Iodine Solution 1.25% w/w [0.125% available iodine] USP
  Single topical administration
  Interventions: Drug: Povidone-Iodine Solution 1.25% w/w [0.125% available iodine] USP

INTERVENTIONS:
Drug: Povidone-Iodine Solution 1.25% w/w [0.125% available iodine] USP — Single topical administration
  Other Names: Halodine Nasal Antiseptic

SUMMARY:
Povidone iodine (PVP-I) is a well-known broad spectrum, resistance free antimicrobial agent that has a long history of safe and effective use. Halodine Nasal Antiseptic is formulated for topical application PVP-I to nasal passages, and has demonstrated effectiveness against SARS-COV-2 in vitro - 99.99% inactivation within 15 seconds. This study will evaluate the ability of Halodine Nasal Antiseptic to impact SARS-CoV-2 in vivo.

DETAILED DESCRIPTION:
This is a multicenter, phase 4 prospective, single-cohort study in adult male and female volunteers hospitalized with COVID-19. Baseline nasopharyngeal swabs will be performed on all individuals. Halodine Nasal Antiseptic will then be applied to the anterior nares. Serial nasopharyngeal samples will then be collected at specified time points after the application. All samples will be tested for SARS-CoV-2 by real-time reverse transcription (rRT)-PCR assay.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with COVID-19
* Positive SARS-CoV-2 (rRT)-PCR within 48 hours of enrollment

Exclusion Criteria:

* Allergies to iodine-containing compounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Nasopharyngeal SARS-CoV-2 Viral Load | 4 hours
  Real-time reverse transcription (rRT)-PCR assay for SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Barone, MD, Study Director — Halodine LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bidra AS, Pelletier JS, Westover JB, Frank S, Brown SM, Tessema B. Rapid In-Vitro Inactivation of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Using Povidone-Iodine Oral Antiseptic Rinse. J Prosthodont. 2020 Jul;29(6):529-533. doi: 10.1111/jopr.13209. Epub 2020 Jun 16. PMID 32511851
- See also: Sponsor's Science Website — https://halodine.com/science/